CLINICAL TRIAL: NCT00887679
Title: Treatment Effects of Escitalopram (Lexapro®) on Generalized Anxiety Disorder, Adherence to Antiretroviral Therapy,Cognition, and Immune Status Among Patients With HIV and AIDS: A 6-week Open-label, Prospective, Pilot Trial.
Brief Title: Treatment Effects of Escitalopram (Lexapro®) on Generalized Anxiety Disorder in Patients With HIV and AIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00011288; LXP-MD-0148
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-03

CONDITIONS: Anxiety Disorders; HIV Infections
Keywords: Escitalopram; Anxiety Disorder; HIV and AIDS; treatment experienced
MeSH Terms: conditions — Anxiety Disorders; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Escitalopram (Experimental): Treatment effects of Escitalopram in Generalized Anxiety Disorder in patients with HIV/AIDS.Open label, rater-blinded, prospective, 6-week trial of escitalopram.Subjects received escitalopram 10-20mg. Escitalopram was started at 10mg per day and augmented weekly in 10mg per day increments, the maximum dose being 20mg per day.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 10-20 mg/day oral of Escitalopram for 6-weeks. Escitalopram flexible dose (10-20 mg/day). A forced escalation schedule of escitalopram was used to titrate it to the maximum tolerated dose. Drug was discontinued at the end of the study.

SUMMARY:
The purpose of this study is to evaluate whether escitalopram is safe, well tolerated, and effective in the treatment of HIV-infected patients with generalized anxiety disorder.

DETAILED DESCRIPTION:
Anxiety disorders are twice as prevalent among HIV-infected patients as they are in the general population. Approximately 25%-40% of HIV-infected patients have anxiety disorders; Generalized Anxiety Disorder, Panic disorder and post-traumatic Stress Disorder being the most frequent. Non-adherence to anti-retroviral medications is commonly seen in patients with HIV with GAD.The role of specific selective serotonin reuptake (SSRIs) in the treatment of HIV-patients with GAD is unclear. Escitalopram has been used in the treatment of GAD in the general population. It has been shown to be safe in HIV-patients with a tolerable side-effect profile. However, whether it can improve GAD in HIV-infected patients has not yet been investigated.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years,
* DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) criteria for Generalized Anxiety Disorder
* confirmed stable HIV disease and attending a HIV treatment program
* stable dose of highly active anti-retroviral therapy for a minimum of 4 weeks
* ability to give informed consent

Exclusion Criteria:

* bipolar disorders, any psychotic disorder
* current major depression
* substance dependence (except nicotine dependence) in the previous 3 months
* currently suicidal or high suicide risk, serious or unstable medical disorders (e.g. uncontrolled hypertension or diabetes)
* any hospitalization for HIV-related illness in the previous 3 months
* any active CNS (central nervous system) CNS opportunistic infection or CNS malignancies related to HIV
* current active treatment for opportunistic infections related to HIV
* any psychotropic drug treatment in the previous 2 weeks before screening
* history of hypersensitivity to escitalopram and/or citalopram
* admission BDI 23
* seizure disorder, traumatic brain injury
* pregnant, nursing mother or planning to get pregnant.
* Concomitant mediations: At least 2-week washout of antidepressant (4 weeks for fluoxetine) or antipsychotic or anti-anxiety medications.
* In the opinion of the investigator the clinical condition precludes participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin A Patkar, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Pence BW, Miller WC, Whetten K, Eron JJ, Gaynes BN. Prevalence of DSM-IV-defined mood, anxiety, and substance use disorders in an HIV clinic in the Southeastern United States. J Acquir Immune Defic Syndr. 2006 Jul;42(3):298-306. doi: 10.1097/01.qai.0000219773.82055.aa. PMID 16639343
- [Background] Tucker JS, Kanouse DE, Miu A, Koegel P, Sullivan G. HIV risk behaviors and their correlates among HIV-positive adults with serious mental illness. AIDS Behav. 2003 Mar;7(1):29-40. doi: 10.1023/a:1022557222690. PMID 14534388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Anxiety disorders in HIV-infected patients from the general population
Groups:
- Escitalopram: Treatment effects of Escitalopram in Generalized Anxiety Disorder in patients with HIV/AIDS.
Period: Overall Study
Arm/Group | Escitalopram
Started | 30
Completed | 20 (20 subjects completed the study.)
Not Completed | 10
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Escitalopram
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Randomization to End of Treatment in Scores on the Hamilton Anxiety Rating Scale (HAM-A)
Description: The HAM-A is administered by an interviewer who asks a series of questions related to symptoms of anxiety. The interviewer then rates the individual on a five-point scale for each of the 14 items. Seven of the items specifically address psychic anxiety and the remaining seven items address somatic anxiety. The total anxiety score ranges from 0 to 56, lower scores are better. Change from randomization to end of treatment in scores on the Hamilton Anxiety Rating Scale (HAM-A)is measured.
Time Frame: baseline and 7 weeks
Population: 3 patients dropped out, 4 patients did not met the criteria, and 3 patients did not show up.
Measure: Mean (Standard Deviation); unit: scores on an anxiety scale
Groups:
- Escitalopram: Treatment effects of Escitalopram in Generalized Anxiety Disorder in patients with HIV/AIDS.Subjects received escitalopram 10-20mg. Escitalopram was started at 10 mg per day and augmented weekly in 10 mg per day increments, the maximum dose being 20 mg per day.
Arm/Group | Escitalopram
Number analyzed (Participants) | 20
scores on an anxiety scale | 21.23 (2.57)

2. Primary Outcome: Changes From Randomization to End of Treatment in Scores on the Beck Depression Inventory
Description: Scoring
  The BDI consist of twenty-one questions about how the subject has been feeling in the last week. Each question has a set of at least four possible answer choices, ranging in intensity as follows:
  (0) I do not feel sad.
  1. I feel sad.
  2. I am sad all the time and I can't snap out of it.
  3. I am so sad or unhappy that I can't stand it.
  A value of 0 to 3 is assigned for each answer and the total score is compared to a key to determine the depression's severity. The standard cut-offs are as follows:[6] 0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.
  Higher total scores indicate more severe depressive symptoms.
Time Frame: baseline and 7 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 20
units on a scale | 27.8 (7.89)

3. Secondary Outcome: Change From Randomization to End of Treatment in Scores for the Clinical Global Impression(CGI-S and CGI-I)
Description: Scale for scoring:
  Clinical Global Impression(CGI-S)
  1. = Normal, no symptoms
  2. = Borderline ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Most extremely ill
  Clinical Global Impression(CGI-I)-improvement since treatment
  1. very much improved
  2. much improved
  3. minimally improved
  4. no change from baseline
  5. minimally worse
  6. much worse
  7. very much worse
Time Frame: baseline and 7 weeks
Population: 3 patients dropped out, 4 patients did not meet criteria, and 3 patients did not show up.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 20
scores on a scale
  Clinical Global Impression (CGI-I) | 1 (0.0)
  Clinical Global Impression (CGI-S) | 2 (1.0)

4. Secondary Outcome: Change From Randomization to End of Treatment for Trail Making Tet (TMT)
Description: Trail Making Test (TMT)Results for TMT are reported as the number of seconds required to complete the task. Higher scores reveal greater impairment.
  Average =29 seconds, Deficient > 78 seconds
Time Frame: baseline to 7 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Escitalopram
Number analyzed (Participants) | 20
seconds | 29.2 (11.23)

5. Secondary Outcome: Changes From Randomization to End of Treatment in Scores on the Mini Mental State Examination (MMSE)
Description: Mini Mental State Examination (MMSE),a low score less than or equal to 23 indicates cognitive impairment and the need for further evaluation; normal cognitive function = 27-30, mild cognitive impairment = 21-26, moderate cognitive impairment = 11-20, and severe cognitive impairment = 0-10. The highest possible score is 30.
Time Frame: baseline and 7 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 20
units on a scale | 0 (0)

6. Secondary Outcome: Changes From Randomization to End of Treatment in Scores on the Sheehan Disability Scores (SDS)
Description: Scoring:
  Participants rate the extent to which work, social life, and home life are impaired by his or her symptoms. A 10 point scale is used where 0= not impaired and 10 is highly impaired indicating. The three aspects of life can be summed up into a single dimensional measure of global functional impairment that indicates 0= not impaired and 30 = highly impaired. Scores of 5 or greater are on any of the three scales are considered significant.
Time Frame: baseline and 7 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 20
units on a scale | 0 (0)

ADVERSE EVENTS:
Arm/Group | Escitalopram
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 21/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=30)
nause (Gastrointestinal disorders) | 7
dizziness (Nervous system disorders) | 4
diarrhea (Gastrointestinal disorders) | 3
dry mouth (Gastrointestinal disorders) | 4
headache (Nervous system disorders) | 1
constipation (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No